CLINICAL TRIAL: NCT03452085
Title: Artificial Saliva in Diabetes Type II: a Randomized Registry Cross Over Study
Brief Title: The Artificial Saliva Spray Reduces Xerostomia in Diabetes Type II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Certmedica International GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IAPSSAPP
Record Dates: First submitted 2018-02-03; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-01

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland; Diabetes Mellitus, Type 2
Keywords: xerostomia; diabetes type II; salivary flow; antioxidant capacity of saliva; aldiamed
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Xerostomia

STUDY DESIGN:
Intervention Model Description: Patients were randomized to two groups, whereas one group starts treatment with AS and the other group starts treatment with TT (control).
  After a wash out phase of 3 days, the patients have to take the other product for also 3 days.
  (e. g. randomized patient takes AS for 3 days, after a wash out period of 3 days he takes TT also for three days.)
Masking Description: The two types of pump-spray had a different bottle design but the bottles were blank with no identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- artificial saliva spray (AS) (Active Comparator): The randomized part of the participants who started first with the artificial saliva spray taking it three times a day for a three days treatment, followed by a wash out phase of 3 days.
  After wash out phase they take for three days the marine water throat spray taking it three times a day for a three days treatment.
  Interventions: Device: artificial saliva spray (AS); Other: maritime throat spray (TT)
- maritime throat spray (TT) (Placebo Comparator): The randomized part of the participants who started first with the marine water throat spray taking it three times a day for a three days treatment, followed by a wash out phase of 3 days.
  After wash out phase they take for three days the artificial saliva spray taking it three times a day for a three days treatment.
  Interventions: Device: artificial saliva spray (AS); Other: maritime throat spray (TT)

INTERVENTIONS:
Device: artificial saliva spray (AS) — cross over design
Other: maritime throat spray (TT) — cross over design

SUMMARY:
In diabetes Type II the xerostomia is a quite frequent symptom. In evaluating the activity of an artificial saliva spray compared to a water gel in patients with Diabetes Type II patients had to follow a three day treatment with each product. Whereas after the first treatment period the two groups had to follow a wash out period of three days before the second treatment period could begin.

The artificial saliva spray reduced the xerostomia and the inflammation or the oral tissue.

DETAILED DESCRIPTION:
In diabetes Type II the xerostomia is a quite frequent symptom. The trial was conducted at a single center. Designed and implementing UNI EN ISO 14155:2012, STROBE statement Version 4 and was in conformity with the guidelines of the Declaration of Helsinki.

The type of study was a randomized, cross over clinical trial to compare two treatments (artificial saliva spray (aldiamed(R) mouth spray) AS vs. (Tonimer(R) Throat Spray) TT .

Twenty one subjects that were part of the epidemiological screening for asymptomatic vascular diseases conducted in the Irwin Lab3 of Spoltore (PE / Italy) The degree of xerostomia for the admission had to be at least > 2 according to a semi-quantal scale (ranging from 0 to 6) and patients already under treatment for xerostomia or with xerostomia score < 2, suffering from obesity, cancer, drug addiction or alcoholism were excluded.

The patients had to follow a three day treatment with each product. Whereas after the first treatment period the two groups had to follow a wash out period of three days before the second treatment period could begin.

The study consisted of a preliminary selection during screening, the measurement of xerostomia and random allocation, first treatment period, wash out period and finally the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

* suffering xerostomia
* degree of xerostomia at least > 2 according to a semiquantal scare ranging from 0 to 6
* diabetes Type II > one year, with stabilized oral hypoglycemic therapy from at least 6 months.
* concomitant chronic diseases pertaining to dyslipidemia, cardiovascular and/or gastrointestinal diseases, and anxiety/depression were accepted provided under adequate therapy since at least 6 months.

Exclusion Criteria:

* under treatment for xerostomia or with xerostomia score < 2
* suffering from obesity (BMI > 30 kg/m2),
* cancer of any type
* drug addiction and alcoholism

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
xerostomia | first day before treatment; change to third day after treatment (day 1+3; 7+9)
  xerostomia was measured according to a semi-quantal visual scale (or VAS; visual analogue scale) ranging from 0 to 6 with intervals of 1 point

SECONDARY OUTCOMES:
stimulated salivary flow | first day before treatment; change to third day after treatment (day 1+3; 7+9)
  Subject was asked to chew a standard square of medical cotton for one minute rolling the cotton in the mouth in order to collect the saliva. The measure of the flow consisted in weighing the cotton before and after the chewing
antioxidant capacity of saliva (SAT test) | first day before treatment; changes to third day after treatment (day 1+3; 7+9)
  The test utilizes the capacity of thiocyanate (SCN) to react with iron (Fe3+) causing the formation of FE((SCN)6)3-.
patients preference for treatment AS or TT | third day after finalization of the treatment period (day 3; 9)
  question in regard to the preference

CONTACTS AND LOCATIONS:
Locations (1):
- Irwin Labs, University of Chieti, Chieti, PE, Italy